CLINICAL TRIAL: NCT07271576
Title: Research on the Role of Phycocyanin in the Prevention, Treatment, and Mechanism of Liver Fibrosis/Cirrhosis
Brief Title: Research on the Protective Effects of Phycocyanin Against Liver Fibrosis and Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0673
Record Dates: First submitted 2025-11-17; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Liver Fibrosis; Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Phycocyanin; maltodextrin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phycocyanin Intervention (Experimental)
  Interventions: Dietary Supplement: phycocyanin
- Maltodextrin Placebo (Placebo Comparator)
  Interventions: Other: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: phycocyanin — Oral phycocyanin formulation treatment, 1.5g/day, for at least 4 weeks (The phycocyanin was provided free of charge by Inner Mongolia Zaihui Shou Bio-engineering Co., Ltd., with company production license number SC12215062400192, executive standard GB 1886.309-2020, food-grade specifications, and batch number E4020250324. All samples used in the clinical study are from the same batch, packaged in opaque aluminum composite bags, 1.5g/bag, and stored frozen).
  Arms: Phycocyanin Intervention
Other: Maltodextrin (Placebo) — This is the placebo control group. The patients will receive the same dosage of maltodextrin for at least 4 weeks.
  Arms: Maltodextrin Placebo

SUMMARY:
This clinical trial aims to determine whether phycocyanin, a natural protein derived from spirulina, can help treat liver fibrosis or cirrhosis in adult patients. The main questions it aims to answer are:

* Can phycocyanin reduce blood levels of liver enzymes (such as ALT and AST) that indicate liver damage?
* Can phycocyanin improve liver stiffness as measured by ultrasound?

Researchers will compare the phycocyanin intervention group with a control group that receives a placebo (a similar-looking maltodextrin supplement without active ingredients) to explore if phycocyanin is more effective in treating liver fibrosis/cirrhosis.

Participants will:

* Take one sachet of either phycocyanin or placebo daily for at least 4 weeks.
* Attend regular clinic appointments (typically every 2-3 months) for routine monitoring of your liver condition, which will include blood and urine tests.
* Provide blood and stool samples once before the treatment and once after the 4-week treatment period.
* Undergo an ultrasound evaluation of liver stiffness.

The study will last approximately 2 years, and the personal information of all patients will be kept strictly confidential.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 75;
* Patients diagnosed with liver fibrosis or cirrhosis;
* Voluntary participation in this study and signing of an informed consent form;
* No acute diseases or significantly worsening symptoms for at least 4 weeks prior to enrollment.

Exclusion Criteria:

* Presence of severe comorbidities;
* Allergy to phycocyanin;
* Patients with a history of severe mental illness that may affect treatment compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-06-04 (Estimated); Study Completion 2027-06-04 (Estimated)

PRIMARY OUTCOMES:
Change in Liver Stiffness Measured by Ultrasound Elastography | Baseline (Day 0) and Post-treatment (Week 4)
  Liver stiffness (kPa) will be quantified using ultrasound elastography to assess fibrosis severity and treatment-related changes.
Change in Serum Alanine Aminotransferase (ALT) Level | Baseline (Day 0) and Post-treatment (Week 4)
  Serum ALT (U/L) will be measured using standard clinical chemistry methods to assess improvement in liver injury following phycocyanin treatment.
Change in Serum Aspartate Aminotransferase (AST) Level | Baseline (Day 0) and Post-treatment (Week 4)
  Serum AST (U/L) will be evaluated to determine liver inflammation status and treatment response.

SECONDARY OUTCOMES:
Gene Expression Changes in Liver Tissue | At the time of liver transplantation surgery (if applicable)
  Liver tissue (~1 cm³) obtained during transplantation (if applicable) will be immediately frozen (-80°C) and analyzed by single-cell or bulk RNA sequencing to explore mechanistic effects of phycocyanin.
Change in Serum IL-6 Concentration | Baseline (Day 0) and Week 4
  Serum IL-6 (pg/mL) will be quantified by immunoassay to evaluate systemic inflammation.
Change in Serum TNF-α Concentration | Baseline (Day 0) and Week 4
  Serum TNF-α (pg/mL) will be measured to assess inflammation associated with liver fibrosis.
Gut Microbiome Composition and Diversity | Baseline (Day 0) and Week 4
  Fecal samples will undergo metagenomic sequencing to evaluate gut microbiome changes, including overall diversity (Shannon Index) and relative abundance (%) of selected microbial taxa (e.g., Bacteroides, Firmicutes).
Change in Serum Metabolite Concentrations Identified by Mass Spectrometry | Baseline (Day 0) and Week 4
  Concentrations (μmol/L) of selected metabolites will be profiled via targeted or untargeted metabolomics to identify metabolic shifts associated with treatment.

OTHER OUTCOMES:
Change in Serum Creatinine Level | Baseline (Day 0) & through study completion, up to 24 months
  Serum creatinine (mg/dL) will be measured to monitor renal safety.
Change in Hemoglobin Level | Baseline (Day 0) & through study completion, up to 24 months
  Hemoglobin (g/dL) will be assessed as part of routine hematology monitoring for safety.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, China